CLINICAL TRIAL: NCT04823702
Title: A Phase I, Open-label, Parallel-group Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of a Single Dose of Aldafermin in Subjects With Impaired Hepatic Function
Brief Title: Study of Aldafermin (NGM282) in Participants With Impaired Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NGM Biopharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 282-HI-104
Record Dates: First submitted 2021-03-26; First posted 2021-04-01 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2021-12

CONDITIONS: Impaired Hepatic Function
MeSH Terms: interventions — aldafermin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Child-Pugh A (Mild Hepatic Impairment) & Healthy Matched (Experimental): Administered by subcutaneous injection
  Interventions: Biological: Aldafermin
- Child-Pugh B (Moderate Hepatic Impairment) & Healthy Matched (Experimental): Administered by subcutaneous injection
  Interventions: Biological: Aldafermin
- Child-Pugh C (Severe Hepatic Impairment) & Healthy Matched (Experimental): Administered by subcutaneous injection
  Interventions: Biological: Aldafermin

INTERVENTIONS:
Biological: Aldafermin — Biological: Aldafermin (NGM282) Subcutaneous Injection
  Other Names: NGM282

SUMMARY:
This is an evaluation of Aldafermin (NGM282) in an open-label, single-dose and parallel group study in participants with Impaired Hepatic Function

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, 18 - 75 years of age, inclusive
2. Able to comprehend and willing to sign an informed consent form (ICF)
3. Willing and able to comply with all study requirements
4. BMI 18 - 40 kg/m2, inclusive at Screening
5. Stable medication regimen - no medication initiation or dose change within 7 days or 5 half-lives (whichever is longer) prior to dosing of the study medication.
6. Non-pregnant, non-lactating females. Female subjects of childbearing potential and male subjects with a female sexual partner of childbearing potential must agree to consistent and adequate birth control. One of the following forms of contraception is required:

   1. Condom
   2. Hormone containing contraceptive
   3. Intrauterine device with a failure rate < 1% per year
   4. Cervical cap or diaphragm with spermicidal agent
   5. Tubal sterilization
   6. Vasectomy in male partner
   7. Sexual abstinence
7. Negative test for drugs of abuse at Screening unless they are currently prescribed
8. Negative human immunodeficiency virus (HIV) antibody screen at Screening

Exclusion Criteria:

1. Any acute disease or condition being treated by medical therapy (prescription or over the counter) known to possibly impact hepatic function
2. History of or recent (< 6 weeks) treatment for a chronic condition with a medication that is known to have hepatotoxic potential.
3. Any significant physical injury or surgical procedure within 6 weeks of Screening
4. Uncontrolled diabetes (hemoglobin A1c [HbA1c] > 9.5%)
5. Uncontrolled hypertension (systolic blood pressure [SBP] > 180 mmHg on ≥ 3 medications of different classes for blood pressure control)
6. Have received any investigational medication within 30 days or 5 half-lives, whichever is longer, prior to study dosing
7. Subjects should not have donated blood within 60 days of study entry or plasma within 7 days of study entry. Subjects must also refrain from blood donation from clinic admission, throughout the study period, and continuing for at least 30 days following the last dose of study medication.
8. Positive urine drug screen at Screening that is not otherwise explained by a permitted concomitant medication
9. History of alcoholism in the 6 months prior to Screening
10. Inadequate peripheral venous access

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of a single dose aldafermin | 4 days
  Maximum observed plasma concentration (Cmax) of aldafermin (Day 1 through Day 4)
Pharmacokinetics of a single dose of aldafermin | 4 days
  Area under the concentration-time curve from time zero extrapolated to infinity (AUC infinity) of aldafermin (Day 1 through Day 4)

SECONDARY OUTCOMES:
Type and frequency of adverse events (Day 1 through Day 11) | 11 days
  Frequency, severity, timing, and/or duration of treatment-emergent adverse events (TEAE) and serious adverse events (SAEs)

OTHER OUTCOMES:
Pharmacodynamics (PD) of biomarker 7-alpha-hydroxy-4-cholesten-3-one (C4) | 6 and 24 hours post dose
  Absolute change from baseline
Pharmacodynamics (PD) of biomarker 7-alpha-hydroxy-4-cholesten-3-one (C4) | 6 and 24 hours post dose
  Percent change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: NGM Study Director, Study Director — NGM Biopharmaceuticals, Inc
Locations (3):
- United States (3):
  - NGM Clinical Study Site 110, Miami, Florida
  - NGM Clinical Study Site 111, Orlando, Florida
  - NGM Clinical Study Site 113, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided